CLINICAL TRIAL: NCT02203435
Title: The Characteristics of the Blue-code Calls; Five Years Survey.
Brief Title: The Patient Characteristics and Mortality of Code Blue Calls
Status: Completed | Type: Observational
Sponsor: Gulsah Karaoren (Other Government)
Responsible Party: Sponsor-Investigator, Gulsah Karaoren, doctor, Umraniye Education and Research Hospital
Organization: Umraniye Education and Research Hospital (Other Government)
Other Study IDs: GK1
Record Dates: First submitted 2014-07-26; First posted 2014-07-29 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Demographics of the Patients Evaluated by Code Blue Call
Keywords: code blue; Cardiopulmonary Resuscitation; APACHE

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aimed to retrospectively examine patients evaluated by the Code Blue team on a Code Blue call in our hospital between 2009 and 2013.

Primary outcome: an examination of the survival rates and demographic data of the patients evaluated as an emergency by a Code Blue call in the period 2009-2013.Secondary outcome: to determine the rates of false Code Blue calls, the clinics giving Code Blue calls and the relationship between the times of Code Blue calls and mortality.Inclusion criteria: patients throughout the whole hospital for whom a Code Blue form was completed and who were evaluated by the Code Blue team on a Code Blue call.

Exclusion criteria: patients who refused treatment

DETAILED DESCRIPTION:
Retrospective examination was made of the Code Blue notification forms which were completed by the anaesthesiologist as Code Blue team leader of the hospital. The age of the patient, gender, diagnosis, the department where admitted, time of Blue Code call, reason for Blue Code call, whether or not the Blue code call was appropriate, whether or not cardiopulmonary resuscitation was administered, if administered, the duration of cardiopulmonary resuscitation, whether or not the patient was postoperative, whether or not the patient had been discharged from the intensive care unit and if so, how many days had passed, the APACHE II score of the patient and expected mortality, were recorded by calculation of the data on thhe Code Blue notification form and in the hospital automated system. Patients were excluded from the study if they had refused treatment or if there was no record of the parameters necessary to calculate the APACHE II score.

ELIGIBILITY:
Inclusion Criteria:

Patients throughout the whole hospital for whom a Code Blue form was completed and who were evaluated by the Code Blue team on a Code Blue call.

Exclusion Criteria:

Patients who refused treatment

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study aimed to retrospectively examine patients evaluated by the Code Blue team on a Code Blue call in our hospital between 2009 and 2013.Retrospective examination was made of the Code Blue notification forms which were completed by the anaesthesiologist as Code Blue team leader of the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
mortality of blue-codes | 5 years
  an examination of the survival rates and demographic data of the patients evaluated as an emergency by a Code Blue call in the period 2009-2013.

SECONDARY OUTCOMES:
the demographics of blue code admissions | 5 years
  to determine the rates of false Code Blue calls, the clinics giving Code Blue calls and the relationship between the times of Code Blue calls and mortality.

OTHER OUTCOMES:
the rate of successful cardiopulmonary resuscitation | 5 years
  the rate of CPR, the apache and saps II expanded values and indication of ICU stay will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Nurten Bakan, assoc prof, Study Director — Istanbul Umraniye Education and Research Hospital
Locations (1):
- Istanbul Umraniye Education and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Grimaldi D, Dumas F, Perier MC, Charpentier J, Varenne O, Zuber B, Vivien B, Pene F, Mira JP, Empana JP, Cariou A. Short- and long-term outcome in elderly patients after out-of-hospital cardiac arrest: a cohort study. Crit Care Med. 2014 Nov;42(11):2350-7. doi: 10.1097/CCM.0000000000000512. PMID 25054671
- [Result] Fecho K, Jackson F, Smith F, Overdyk FJ. In-hospital resuscitation: opioids and other factors influencing survival. Ther Clin Risk Manag. 2009;5:961-8. doi: 10.2147/tcrm.s8121. Epub 2009 Dec 29. PMID 20057895
- [Result] Yang J, Howell MD. Commentary: Is the glass half empty? Code blue training in the modern era. Acad Med. 2011 Jun;86(6):680-3. doi: 10.1097/ACM.0b013e318217e969. PMID 21613890